CLINICAL TRIAL: NCT02627690
Title: Nephrologic Prognosis 10 Years After Diabetes Cell Therapy
Acronym: PRONOCELDIAB
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_28; 2014-A00141-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-02-05; First posted 2015-12-11 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Islet Transplantation
MeSH Terms: interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Islet transplanted: patients who underwent islet transplantation
  Interventions: Other: islet transplanted
- non islet transplanted: patients who refused or were non selected for islet transplantation for a non nephrologic reason
  Interventions: Other: non islet transplanted

INTERVENTIONS:
Other: islet transplanted — islet transplantation
  Other Names: Islet transplantation
  Groups: Islet transplanted
Other: non islet transplanted — no islet transplantation (for a non nephrologic reason)
  Other Names: no islet transplantation
  Groups: non islet transplanted

SUMMARY:
Islet transplantation for type 1 diabetes results are still improving, and actually Insulin-independence with normal HbA1c is obtained in 50% of patients after 5 years, 80% of c-peptide positive patients. In addition to the need of 2 or 3 surgical or radiological interventions to inject islets, an immunosuppressive regimen is needed, which can be deleterious, particularly on kidneys. Moreover, long term beneficial effects of islet transplantation on stabilization or prevention of macro and micro vascular complications of diabetes has not been evaluated. In a preliminary work, it was observed a stabilisation or improvement of microvascular complications when compared to pre-transplant data.

The aim of this study is to compare the evolution of diabetes complications, especially nephrologic, 10 years after islet transplantation and to compare it to patients with a brittle diabetes, 10 years after evaluation for islet transplantation, finally not performed.

This case-control study will evaluate nephrologic parameters (creatinine, MDRD creatinine clearance, microalbuminuria, proteinuria) and other micro and macro-vascular complications of type 1 diabetes) before islet transplantation and 10 years after the transplantation or after the first evaluation in patients who finally did not underwent islet transplantation for various non nephrologic reasons

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patients, with or without previous renal transplantation who benefit at least 5 years before the inclusion of clinical evaluation in order to perform an islet transplantation
* Who either benefit of islet transplantation or did not and treated with optimized insulin therapy

Exclusion Criteria:

* C-peptide positive diabetes
* Type 1 diabetic patient non-grafted of islets due to albuminuria> 300mg / 24h or MDRD <50 ml / min during the pre-transplant evaluation (exclusion criterion for islet transplantation)
* Patients that can not receive clear information
* Refusal to sign the consent
* Psychiatric Pathology
* Participation in another study excluding the possibility of participating in another protocol.
* Pregnant or breast feeding women
* Patients under guardianship, persons deprived of freedom
* Lack of coverage by the social security system

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering of type 1 diabetes since at least 10 years
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Modification of Diet in Renal Disease (MDRD) | At 10 years
  measure the difference of Modification of Diet in Renal Disease (MDRD) between the two groups according to the presence or absence of an islet transplant.

SECONDARY OUTCOMES:
number of cardiovascular events | At 10 years
number of deaths | At 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine VANTYGHEM, MD, PhD, Principal Investigator — Lille University Hospital
Locations (1):
- Lille University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: No